CLINICAL TRIAL: NCT05197088
Title: Medication Facilitated Ureteral Access Sheath Deployment During Ureteroscopy: the Impact of One Week of Pre-operative Tamsulosin
Brief Title: Tamsulosin Assisted Ureteral Access Sheath Insertion
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Sundaram Palaniappan, Dr, Sengkang General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/2156
Record Dates: First submitted 2022-01-09; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Renal Stone; Retrograde Intrarenal Surgery; Urolithiasis
MeSH Terms: conditions — Nephrolithiasis; Urolithiasis | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 week of tamsulosin (Experimental): 1 week of tamsulosin tablet 400mcg once a night
  Interventions: Drug: Tamsulosin
- no additional medication (No Intervention)

INTERVENTIONS:
Drug: Tamsulosin — 1 week of tamsulosin
  Arms: 1 week of tamsulosin

SUMMARY:
Aim is to study if 1 week of pre operative tamsulosin would enable easier insertion of ureteral access sheath in primary retrograde intrarenal surgery for renal stone disease

ELIGIBILITY:
Inclusion Criteria:

* renal stone undergoing retrograde intrarenal surgery

Exclusion Criteria:

* not on tamsulosin or other alpha blockers regularly
* ureteral stricture
* concurrent ureteric stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01-09 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
successful insertion of ureteral access sheath to the upper ureter (above the level of SI joint on fluoroscopy) | during operation

SECONDARY OUTCOMES:
grade of ureteric injury after ureteral access sheath removal | during operation
post operative complications | 3 months
stone free rate | 3 months
need for additional procedures | 3 months

IPD SHARING:
Plan to Share IPD: No